CLINICAL TRIAL: NCT01774682
Title: Does the Sleeve Gastrectomy Improve the Kinematics of Obese Patients Perambulation ?
Brief Title: Kinematics of Obese Patients Perambulation
Acronym: MARCHOBESE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI11-PR-VERHAEGHE; 2012-A00153-40 (Other: ANSM)
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Morbid Obesity; Surgical Management by Laparoscopic Sleeve Gastrectomy
Keywords: obesity; surgery
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 6-minute walk test (Other): the 6-minute walk test is performed for each patient prior to the surgery and 6 months after by a specialist.
  Interventions: Procedure: 6-minute walk test

INTERVENTIONS:
Procedure: 6-minute walk test — the test corresponds to that defined by Abdel Kafi et al in 2005

SUMMARY:
The aim of this study is to evaluate the consequences of sleeve gastrectomy on functional parameters of patients perambulation.

DETAILED DESCRIPTION:
Laparoscopic Sleeve gastrectomy is the standard surgical procedure for the treatment of obese patients. Even the surgery is well described, there is no available study about its influence on the functional parameters of patients perambulation.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 40 and 60 kg/m2 or BMI > 35 kg/m2 with at least one comorbidity
* no weight loss
* between 18 and 65 years old
* history of obesity > 5 ans

Exclusion Criteria:

* history of bariatric surgery
* major cardiac insufficiency
* pregnancy or breastfeeding
* no social welfare

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
6-minute walk test | 6 months after the surgery
  the value of this test is obtained by the difference between the 6-minute walk test performed before the surgery and the 6-minute walk test performed 6 months after the surgery

SECONDARY OUTCOMES:
quality of life | 6 months after the surgery
  the quality of life is evaluated by the SF36 questionnaire which is performed before the surgery and 6 months after.
BAROS score | 6 months after the surgery
  the baros score is evaluated by the surgeon during the consultation 6 months after the surgery
quality of life with the Mooreheald-Ardelt questionnaire | 6 months after the surgery
  the Mooreheald-Ardelt questionnaire is completed by the patient during the consultation 6 months after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: abdennaceur dhahri, MD, Principal Investigator — CHU Amiens
Locations (1):
- Chu Amiens, Amiens, France

REFERENCES:
- [Background] Rebibo L, Fuks D, Verhaeghe P, Deguines JB, Dhahri A, Regimbeau JM. Repeat sleeve gastrectomy compared with primary sleeve gastrectomy: a single-center, matched case study. Obes Surg. 2012 Dec;22(12):1909-15. doi: 10.1007/s11695-012-0779-9. PMID 23001573
- [Background] Rebibo L, Dhahri A, Verhaeghe P, Regimbeau JM. Early gastric fistula after laparoscopic sleeve gastrectomy: surgical management. J Visc Surg. 2012 Oct;149(5):e319-24. doi: 10.1016/j.jviscsurg.2012.07.004. Epub 2012 Aug 9. No abstract available. PMID 22884227
- [Background] Pequignot A, Dhahri A, Verhaeghe P, Desailloud R, Lalau JD, Regimbeau JM. Efficiency of laparoscopic sleeve gastrectomy on metabolic syndrome disorders: two years results. J Visc Surg. 2012 Oct;149(5):e350-5. doi: 10.1016/j.jviscsurg.2012.06.005. Epub 2012 Jul 17. PMID 22809752
- [Background] Rebibo L, Mensah E, Verhaeghe P, Dhahri A, Cosse C, Diouf M, Regimbeau JM. Simultaneous gastric band removal and sleeve gastrectomy: a comparison with front-line sleeve gastrectomy. Obes Surg. 2012 Sep;22(9):1420-6. doi: 10.1007/s11695-012-0689-x. PMID 22790710
- [Background] Dhahri A, Verhaeghe P, Hajji H, Fuks D, Badaoui R, Deguines JB, Regimbeau JM. Sleeve gastrectomy: technique and results. J Visc Surg. 2010 Oct;147(5 Suppl):e39-46. doi: 10.1016/j.jviscsurg.2010.08.016. No abstract available. PMID 20971049
- [Result] Rebibo L, Verhaeghe P, Tasseel-Ponche S, Cosse C, Marechal V, Dhahri A, Doutrellot PL, Regimbeau JM. Does sleeve gastrectomy improve the gait parameters of obese patients? Surg Obes Relat Dis. 2016 Sep-Oct;12(8):1474-1481. doi: 10.1016/j.soard.2016.03.023. Epub 2016 Mar 25. PMID 27387694